CLINICAL TRIAL: NCT04677088
Title: Phase I Study of T Cell Receptor-Redirected T Cells With Recurrent HBV Treatment in Patients-Related Hepatocellular Carcinoma in Post Liver Transplantation
Brief Title: TCR-Redirected T Cell Treatment in Patients With Recurrent HBV-related Hepatocellular Carcinoma Post Liver Transplantation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xiaoshun He (Other)
Collaborators: Lion TCR Pte. Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Xiaoshun He, MD., First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTCR-HCC-2-2
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Recurrent Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HBV/ TCR T cell infusion (Experimental): Autologous T cells with HBV antigen-specific TCR
  Interventions: Biological: TCR-T cells

INTERVENTIONS:
Biological: TCR-T cells — Patients will receive 1 x 10^4 cells/kg to 5 x 10^6 cells/kg bodyweight of TCR redirected T cells by IV infusion.

SUMMARY:
This is a single-arm and open-label study to assess the safety, tolerability and primary efficacy of the HBV specific T cell receptor (HBV/TCR) redirected T cell in patients with recurrent Hepatitis B virus (HBV) related hepatocellular carcinoma post liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis as hepatocellular carcinoma (HCC).
2. Recurrent locally advanced and/or metastatic hepatocellular carcinoma (HCC) post liver transplantation.
3. Seropositive for hepatitis B surface antigen, or presence of HBV DNA or HBV RNA.
4. HLA profile matching with HLA-class I restriction element of the available T cell receptors.
5. ECOG performance status ≤ 2.
6. Laboratory criteria:

   1. Liver function: ALT and AST ≤ 5 of upper limit of normal (ULN), TBIL ≤ 3 x ULN.
   2. Neutrophil cell number ≥1.5×10^9/L.
   3. Platelet count ≥100×10^9/L.
7. Ability to provide informed consent.
8. Willing and able to comply with all study procedures.

Exclusion Criteria:

1. Second primary malignancy that is clinically detectable at the time of consideration for study enrolment.
2. Likelihood to require steroid treatment during the period of the clinical trial.
3. Lack of peripheral venous or central venous access or any condition that would interfere with drug administration or collection of study samples.
4. Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
5. Administration of any other cell therapy, including NK, CIK, DC, CTL, CAR- T, stem cells or combined therapy of the kind within 28 days prior to start of treatment.
6. Any condition that is unstable or which could jeopardise the safety of the patient and his/her compliance in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation of the TCR-T treatment | Start of Treatment until 28 days post last dose
  Incidence of adverse events/serious adverse events

SECONDARY OUTCOMES:
Overall Response Rate | Start of treatment until disease progression, and subsequent follow up up to 24 months post treatment.
  Tumour assessment will be according to RECIST v1.1. This is based on percentage of participants with Complete Response (CR) and Partial Response (PR) according to RECIST v1.1 from baseline.
Progression-free survival (PFS) | Start of treatment until disease progression, and at 6-month and 1-year.
  1-year PFS is measured by the number of patients with stable disease after 1 year, using RECIST v1.1.
Overall survival (OS) | Start of treatment until disease progression, and at 6-month and 1-year.
  OS is defined as the time from randomisation until death by any cause. Participants will be followed up for survival follow up for two years.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun-Yat Sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Tan AT, Yang N, Lee Krishnamoorthy T, Oei V, Chua A, Zhao X, Tan HS, Chia A, Le Bert N, Low D, Tan HK, Kumar R, Irani FG, Ho ZZ, Zhang Q, Guccione E, Wai LE, Koh S, Hwang W, Chow WC, Bertoletti A. Use of Expression Profiles of HBV-DNA Integrated Into Genomes of Hepatocellular Carcinoma Cells to Select T Cells for Immunotherapy. Gastroenterology. 2019 May;156(6):1862-1876.e9. doi: 10.1053/j.gastro.2019.01.251. Epub 2019 Jan 31. PMID 30711630
- [Background] Qasim W, Brunetto M, Gehring AJ, Xue SA, Schurich A, Khakpoor A, Zhan H, Ciccorossi P, Gilmour K, Cavallone D, Moriconi F, Farzhenah F, Mazzoni A, Chan L, Morris E, Thrasher A, Maini MK, Bonino F, Stauss H, Bertoletti A. Immunotherapy of HCC metastases with autologous T cell receptor redirected T cells, targeting HBsAg in a liver transplant patient. J Hepatol. 2015 Feb;62(2):486-91. doi: 10.1016/j.jhep.2014.10.001. Epub 2014 Oct 13. PMID 25308176
- [Background] Gehring AJ, Xue SA, Ho ZZ, Teoh D, Ruedl C, Chia A, Koh S, Lim SG, Maini MK, Stauss H, Bertoletti A. Engineering virus-specific T cells that target HBV infected hepatocytes and hepatocellular carcinoma cell lines. J Hepatol. 2011 Jul;55(1):103-10. doi: 10.1016/j.jhep.2010.10.025. Epub 2010 Nov 23. PMID 21145860
- [Background] Koh S, Shimasaki N, Suwanarusk R, Ho ZZ, Chia A, Banu N, Howland SW, Ong AS, Gehring AJ, Stauss H, Renia L, Sallberg M, Campana D, Bertoletti A. A practical approach to immunotherapy of hepatocellular carcinoma using T cells redirected against hepatitis B virus. Mol Ther Nucleic Acids. 2013 Aug 13;2(8):e114. doi: 10.1038/mtna.2013.43. PMID 23941866